CLINICAL TRIAL: NCT02415946
Title: Efficacy of a Novel Simplified, Minimally-invasive Procedure for Sinus Floor Elevation in the Atrophic Posterior Maxilla: a Multicenter, Randomized Study
Brief Title: Sinus Lift: Saving Time and Reducing Morbidity
Acronym: SmartLiftRER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Roberto Farina, Full-Time Researcher, Chair of Oral Implantology, University of Ferrara, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRUA1GR-2013-00000168
Record Dates: First submitted 2014-12-02; First posted 2015-04-14 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Tooth Loss; Bone Atrophy
Keywords: regenerative medicine; bone substitutes; sinus floor augmentation
MeSH Terms: conditions — Tooth Loss | interventions — Sinus Floor Augmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sinus floor augmentation (lateral) (Active Comparator): Maxillary sinus floor elevation using a lateral approach
  Interventions: Procedure: Sinus floor augmentation (lateral)
- Sinus floor augmentation (transcrestal) (Experimental): Maxillary sinus floor elevation using a transcrestal approach (Smart Lift technique; Trombelli et al. 2008)
  Interventions: Procedure: Sinus floor augmentation (transcrestal)

INTERVENTIONS:
Procedure: Sinus floor augmentation (lateral)
  Arms: Sinus floor augmentation (lateral)
Procedure: Sinus floor augmentation (transcrestal)
  Arms: Sinus floor augmentation (transcrestal)

SUMMARY:
BACKGROUND Tooth loss impairs the OHRQoL. Dental implants have expanded treatment options of edentulous patients and improved their OHRQoL, however, in the posterior maxillary sextants the possibility to place implants of desired length and diameter could be limited. lSFE and tSFE represent two surgical options to vertically enhance the available bone in the edentulous posterior maxilla. Invasivity, relevant postoperative discomfort, high costs, and long times needed for the finalization of the prosthetic rehabilitation, however, strongly limit the indications of lSFE and support the need for less traumatic procedures with similar clinical effectiveness and reduced morbidity. In 2008, the investigators proposed a user-friendly, safe, predictable and effective minimally-invasive procedure for tSFE, namely the Smart Lift technique.

AIMS/OBJECTIVES The general aim of the present project is to validate the Smart Lift technique as a simplified and minimally-invasive procedure for the implant-supported rehabilitation of patients with edentulous, atrophic maxillary posterior sextants.

METHODS In a multicenter RCT study design, the reconstructive (clinical) and patient-centered outcomes of tSFE performed according to the Smart Lift technique will be compared with those of conventional lSFE.

EXPECTED RESULTS The Smart Lift technique should allow for a significant reduction of treatment time, post-surgery complications and costs and an increase in the satisfaction perceived by the edentulous patient with implant-supported rehabilitation, while maintaining a clinical efficacy as well as a similar or lower morbidity and discomfort when compared to lSFE. In other words, the investigators expect that more favorable risk-benefit and cost-utility ratio, as well as a better performance in terms of pain, comfort, physical, social and psychological effects of oral health, and issues concerning the OHRQoL, will be observed for the Smart Lift technique compared to lSFE.

List of Acronyms (in alphabetical order) OHRQoL: Oral Health - Related Quality of Life lSFE: sinus floor elevation with a lateral approach RCT: randomized controlled trial tSFE: sinus floor elevation with transcrestal approach

ELIGIBILITY:
Inclusion Criteria:

Patient-specific

* age≥ 21 years;
* good physical status (ASA1 and ASA2 according to Physical Status Classification System) (American Society of Anesthesiologists);
* systemic and local conditions compatible with implant placement and sinus floor elevation procedures;
* indication to a fixed, implant-supported prosthetic rehabilitation with sinus floor elevation as part of the comprehensive oral rehabilitation plan;
* patient willing and fully capable to comply with the study protocol.

Site-specific For a site to be considered as experimental (and thus included for analysis), the following criteria must be fulfilled:

* at least 6 months elapsed from tooth/teeth loss;
* residual bone height (as radiographically assessed) ≥3 mm and ≤6 mm;
* receiving an implant 3.5 ÷ 5 mm wide, ≥ 8 mm long and at least 5 mm longer than the residual bone height.

Exclusion Criteria:

* current heavy smoking (≥ 20 cigarettes/day for ≥ 6 months prior to and at the time of the surgical procedure);
* untreated periodontal disease prior to implant placement;
* history of radiation therapy in the head and neck area;
* history of chemotherapy;
* systemic disease or conditions with a documented effect on bone metabolism and/or osseous healing;
* past (within 6 months prior to enrollment in the study) or current treatment with any medication with a documented effect on bone metabolism and/or osseous healing;
* physical or mental handicap that can interfere with adherence to the study procedures and adequate hygienic compliance;
* documented allergy to dental materials involved in the experimental protocol;
* pregnancy or lactation;
* history of drug or alcohol abuse.

Moreover, participants will be exited from the study immediately upon:

* request to withdraw from further participation;
* development of acute dental, peri-implant or oral conditions requiring treatment;
* development of conditions conflicting with the exclusion criteria listed above;
* failure to comply with study instructions/requirements.

Site-specific

* presence of endodontic lesions at teeth adjacent to the implant site;
* previous bone augmentation/preservation procedures at the designated implant areas;
* diagnosis of maxillary sinusitis at the experimental quadrant;
* need for concomitant lateral/vertical bone reconstructive procedures other than maxillary sinus floor elevation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Vertical extent of sinus lift | week +48
  At each observation interval, the vertical extent of sinus lift will be measured as the distance (in mm) between the sinus floor and the most apical portion of the radiopaque area in the mid CT/CBCT section including the implant.

SECONDARY OUTCOMES:
Implant survival | week +48
  At each observation interval, implant survival will be recorded as the persistence of the implant in the oral cavity with absence of mobility (defined as the absence of vertical, lateral and rotational movements of the implant). When evaluating multiple implants splinted by prosthetic restorations, all implants supporting the prosthesis will be considered as failed or survived if the prosthesis is mobile or not mobile, respectively.
Type and incidence of surgical and post-surgical complications | week +48
  The incidence of membrane perforation will be evaluated by the Valsalva maneuver (for tSFE) or visually (for lSFE). Other surgical or post-surgical complications associated with the sinus lift procedure, including Benign Paroxysmal Positional Vertigo (BPPV), post-operative infection, post-operative haemorrhage, nasal bleeding, blocked nose, either assessed by the operator or reported by the patient, will be also recorded.
Level of post-operative pain | week +2
  The level of pain perceived by the patient (VASpain) will be recorded daily (evening) for 14 days following surgery on a 100-mm visual analogue scale (VAS) (ranging from "0 - no pain" to "100 - intolerable pain").
type and dosage of post-surgery medications | week +2
  The patient will self-report the dosage of rescue anti-inflammatory drug (i.e. number of ibuprofen 600 mg tablets) assumed from the 1st to the 14th postoperative day, as well as the assumption of other types of drugs (e.g. antibiotics).
Costs arised from the realization of the surgical procedure and during the postoperative period | week +48
  Costs arised (i) from the realization of the surgical procedure (e.g., pre-operative exams, materials), and (ii) during the postoperative period (e.g., patient post-surgical monitoring, management of post-surgical complications, and limitations in daily activities caused by surgery) will be evaluated for each patient.
  Rather than with monetary units, costs will be compared between treatment groups using tSFE/lSFE ratios.
radiographic height of the graft over the implant apex | week +48
  The height of the graft apical to the implant apex will be measured as the distance (in mm) occupied by a radiopaque area between the implant apex and the sinus floor as assessed at the mid portion of the implant on the mid CT/CBCT section including the implant.
General health-related quality of life as assessed by the Short Form Health Survey (SF-36) questionnaire | day 0, week +48
  A validated, self-administered questionnaire will be used to assess the general health - related quality of life (GHrQoL) immediately before surgery and at week +48. To assess GHrQoL, the Short Form health survey (SF-36) questionnaire (Ware & Sherbourne 1992) will be used.
Oral health-related quality of life as assessed by the Oral Health Impact Profile (OHIP-20) questionnaire | day 0, week +48
  A validated, self-administered questionnaire will be used to assess the oral health - related quality of life (OHrQoL) immediately before surgery and at week +48. To assess OHrQoL, the Oral Health Impact Profile (OHIP)-20 questionnaire (Allen & Locker 2002, Awad et al. 2003) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Farina, Researcher, Principal Investigator — Research Centre for the Study of Periodontal and Peri-implant Diseases, University of Ferrara, Italy
Locations (2):
- Italy (2):
  - University-Hospital, Ferrara
  - University-Hospital, Modena

REFERENCES:
- [Derived] Farina R, Simonelli A, Franceschetti G, Minenna L, Schincaglia GP, Riccardi O, Trombelli L. Peri-implant tissue conditions following transcrestal and lateral sinus floor elevation: 3-year results of a bi-center, randomized trial. Clin Oral Investig. 2022 May;26(5):3975-3986. doi: 10.1007/s00784-021-04364-y. Epub 2022 Jan 10. PMID 35013782
- [Derived] Farina R, Franceschetti G, Travaglini D, Consolo U, Minenna L, Schincaglia GP, Riccardi O, Bandieri A, Maietti E, Trombelli L. Radiographic outcomes of transcrestal and lateral sinus floor elevation: One-year results of a bi-center, parallel-arm randomized trial. Clin Oral Implants Res. 2019 Sep;30(9):910-919. doi: 10.1111/clr.13497. Epub 2019 Jul 10. PMID 31240743
- [Derived] Farina R, Franceschetti G, Travaglini D, Consolo U, Minenna L, Schincaglia GP, Riccardi O, Bandieri A, Maietti E, Trombelli L. Morbidity following transcrestal and lateral sinus floor elevation: A randomized trial. J Clin Periodontol. 2018 Sep;45(9):1128-1139. doi: 10.1111/jcpe.12985. Epub 2018 Aug 3. PMID 29992594